CLINICAL TRIAL: NCT05155943
Title: A Prospective, Non-randomized, Single-arm Study to Evaluate the Safety and Performance of the KALPA X™ Mapping, Imaging, and Navigation Device in Patients Undergoing Left Atrial Appendage Closure (LAAC)
Brief Title: K2 Medical KALPA X™ Mapping, Imaging and Navigation Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The intended population has been updated
Sponsor: Cara Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KADILAC 1.0
Record Dates: First submitted 2021-09-20; First posted 2021-12-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2021-09

CONDITIONS: Left Atrial Appendage Aneurysm
Keywords: LAA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KALPA X (Experimental): The KALPA™ and KALPA X™ systems will be used during the performance of the LAAC procedure that is performed using customary and conventional tools and imaging technologies as currently performed in the participating center.
  Interventions: Device: KALPA X™

INTERVENTIONS:
Device: KALPA X™ — Before and after a transseptal puncture, the right atrium (RA), left atrial appendage (LAA), and left upper superior pulmonary vein (LUSPV) will be mapped using the KALPA™ system (WS Software ver. 1.0.229-0 Source control ID: 65f1dbf7) in combination with a commercially available catheter. Subjects will then undergo LAAC as per routine clinical care. The entire LAAC procedure will be conducted as customary practice using standard and approved off-the-shelf equipment (body surface electrodes, catheters, etc.) the operator will be blinded to the KALPA™ and KALPA X™ system information.

SUMMARY:
This prospective, multi-center, non-randomized, single-blinded, open-label, single-arm, comparator study will enroll up to 100 eligible subjects from multiple sites undergoing LAAC procedure to evaluate the safety and performance of the KALPA™ mapping, imaging and navigation device in patients undergoing Left Atrial Appendage Closure (LAAC).

DETAILED DESCRIPTION:
All subjects will undergo pre-procedural cardiac computed tomography angiography (CCTA) no more than 1 year prior to the performance of the LAAC procedure to evaluate left atrial appendage (LAA) anatomy. Before and after a transseptal puncture, the right atrium (RA), left atrial appendage (LAA), and left upper superior pulmonary vein (LUSPV) will be mapped using the KALPA™ system in combination with a commercially available catheter. Subjects will then undergo LAAC as per routine clinical care. Following implantation of the LAAC device, subjects will be assessed for the peri-device leak (PDL) with a transesophageal echocardiogram (TEE) as well as PDL assessment using the KALPA X™ system (the operator will be blinded to KALPA X™ PDL reading). The entire LAAC procedure will be conducted as customary practice using standard and approved off-the-shelf equipment (body surface electrodes, catheters, etc.) the operator will be blinded to the KALPA™ and KALPA X™ system information. The physician will neither use nor rely on any of the KALPA™ or KALPA X™system output for clinical decision-making.

All patients will then undergo cardiac computed tomography angiography (CCTA) and TEE at 45 days following the index LAAC procedure to assess residual PDL. Intra-procedure PDL post-LAAC assessed by KALPA X™ will be compared to the detection of PDL by TEE. The value of PDL as measured by TEE compared to KALPA X™ at the time of the index LAAC procedure in predicting PDL at 45 days post-LAAC as assessed by CCTA will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥ 18 years of age.
2. The patient meets indications for LAAC procedure.
3. LAAC will be performed using the AMPLATZER Amulet device (AMPLATZER™ Amulet™ LAA Occluder, Abbott Vascular, Santa Clara, CA, USA), or, WATCHMAN (WATCHMAN™ LAAC Device or WATCHMAN FLX™ LAAC Device, Boston Scientific Marlborough, MA, USA) devices, or LAmbre LAA closure system (Lifetech Scientific Co, Ltd, Shenzhen, China), or any other LAA closure device commercially available at the discretion of the principal investigator.
4. The patient is willing to comply with specified follow-up evaluations.
5. The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics Committee (EC)

Exclusion Criteria:

1. Pregnant or nursing subjects. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to index procedure per site standard test.
2. Patients with known atrial septal defect or atrial septal repair or closure device that would preclude transseptal puncture for LAAC.
3. Patients who have a planned treatment with any other investigational device or procedure during the study period.
4. Contraindications to transesophageal echocardiography (TEE), including recent esophageal or gastric surgery (within 6 months), esophageal obstruction (stricture or tumor), depressed respiratory function, active upper gastrointestinal bleeding, perforate viscous (known or suspected), or uncooperative patient.
5. Contraindications to cardiac computed tomography angiography (CCTA) including pregnancy or hypersensitivity to iodinated contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with KALPA X™ device-related adverse events | Up to 24 hours
  Safety of using KALPA X™ during a cardiac procedure, specifically the safety of using KALPA™ during the LAAC procedure, by collecting the records of device related AE's
LAA maximum diameter and perimeter assessed by KALPATM compared to cardiac CT | Up to 24 hours
  Measures of LAA maximum diameter and perimeter obtained by KALPATM performed during the LAAC procedure will be compared to these measurements obtained by the pre-procedure cardiac CT
Multi-Modality Assessment of Immediate Post-LAAC Peri-Device Leak (PDL) by TEE and KALPA X™ | Up to 24 hours
  PDL measured by KALPA X™ (defined below) will be assessed compare to the PDL detected by TEE

SECONDARY OUTCOMES:
Follow-up PDL | Up to 45 days
  The predictive power of intra-procedural TEE and KALPA X™ for the detection of PDL will be compared to 45 day post-LAAC PDL as detected by TEE and CCTA

CONTACTS AND LOCATIONS:
Overall Officials: Helena Grinberg, PhD, Study Director — K2 Medical
Locations (2):
- Policlinico San Donato, Milan, Italy
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided